CLINICAL TRIAL: NCT06884514
Title: Acute Effects of MDMA Co-administration on the Response to Psilocybin in Healthy Subjects
Acronym: MDMA-Psilo
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BASEC 2024-00893
Record Dates: First submitted 2025-01-31; First posted 2025-03-19 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Healthy
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, 4-period cross-over design with three active substance conditions and placebo:
  1. 20 mg Psilocybin + MDMA placebo
  2. Psilocybin placebo + 100 mg MDMA
  3. 20 mg Psilocybin + 100 mg MDMA
  4. Psilocybin placebo + MDMA placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 20 mg Psilocybin + MDMA placebo (Experimental): 20 mg Psilocybin + MDMA placebo
  Interventions: Drug: Psilocybin; Drug: 3,4-Methylenedioxymethamphetamine placebo
- Psilocybin placebo + 100 mg MDMA (Experimental): Psilocybin placebo + 100 mg MDMA
  Interventions: Drug: 3,4-Methylenedioxymethamphetamine; Drug: Psilocybin placebo
- 20 mg Psilocybin + 100 mg MDMA (Experimental): 20 mg Psilocybin + 100 mg MDMA
  Interventions: Drug: Psilocybin; Drug: 3,4-Methylenedioxymethamphetamine
- Psilocybin placebo + MDMA placebo (Placebo Comparator): Psilocybin placebo + MDMA placebo
  Interventions: Drug: Psilocybin placebo; Drug: 3,4-Methylenedioxymethamphetamine placebo

INTERVENTIONS:
Drug: Psilocybin — A moderate dose of 20 mg psilocybin will be administered.
  Arms: 20 mg Psilocybin + 100 mg MDMA; 20 mg Psilocybin + MDMA placebo
Drug: 3,4-Methylenedioxymethamphetamine — A moderate dose of 100 mg MDMA will be administered.
  Arms: 20 mg Psilocybin + 100 mg MDMA; Psilocybin placebo + 100 mg MDMA
Drug: Psilocybin placebo — Mannitol capsules instead of capsules containing psilocybin.
  Arms: Psilocybin placebo + 100 mg MDMA; Psilocybin placebo + MDMA placebo
Drug: 3,4-Methylenedioxymethamphetamine placebo — Mannitol capsules instead of capsules containing MDMA.
  Arms: 20 mg Psilocybin + MDMA placebo; Psilocybin placebo + MDMA placebo

SUMMARY:
The acute subjective effects of serotonin (5-HT)2A receptor stimulation with psilocybin in humans are mostly positive. However, negative effects such as anxiety, paranoid thinking, or loss of trust towards other people are common effects, depending on the dose administered, the personality traits of the person consuming it (set), or the environment in which psilocybin is taken (setting). Negative psychedelic effects may cause acute distress to the subject and acute anxiety has been linked to less favorable long-term outcomes in patients experimentally treated with psilocybin or similar substances for the treatment of depression. The 5-HT and oxytocin releaser 3,4-methylenedioxymethamphetamine (MDMA) reliably induces positive mood, euphoria, comfort, empathy, and feelings of trust. If administered in combination with psilocybin, MDMA may increase positive subjective drug effects including positive mood, empathy, and trust and reduce negative emotions and anxiety associated with psilocybin and overall produce a more positive over negative experience. The present study will assess subjective and autonomic effects of psilocybin alone and in combination with MDMA.

DETAILED DESCRIPTION:
Psilocybin is a classic serotonergic psychedelic. Clinically, the acute effects of psilocybin last shorter than those of lysergic acid diethylamide (LSD) but are qualitatively very similar. Currently, psilocybin is the most investigated psychedelic substance among the classic psychedelics including LSD, psilocybin, mescaline, and dimethyltryptamine (DMT). Psilocybin is capable of inducing exceptional subjective effects such as a dream-like alteration of consciousness, affective changes, psychological insight, visual imagery, pseudo-hallucinations and ego-dissolution. The acute subjective effects elicited by psilocybin are mostly positive in humans. However, psychedelic substances like psilocybin may also cause unpleasant subjective effects like negative thoughts, rumination, anxiety, panic, paranoia, loss of trust towards other people and perceived loss of control, depending on the dose of psilocybin used, the personality traits of the person consuming it (i.e. 'set'), the environment in which it is consumed (i.e. 'setting'), and other factors. Acute negative psychological effects are considered the main risk of psychedelic substance use in humans. Inducing an overall positive acute response to the psychedelic is critical because several studies showed that a more positive experience is predictive of a greater therapeutic long-term effect of the psychedelic. The present study uses 3,4-methylenedioxymethamphetamine (MDMA) as a pharmacological tool to optimize the effects of psilocybin by inducing positive mood. MDMA is an amphetamine derivative which, unlike prototypical amphetamines, predominantly enhances serotonergic neurotransmission via release of 5-HT through the serotonin transporter (SERT). Furthermore, MDMA is known to trigger oxytocin release which may contribute to its effects to increase trust, prosociality, and enhanced empathy. The state of well-being induced by MDMA including increased activation and emotional excitation is known to be associated with a better response to psychedelics. Due to its psychological profile, MDMA could be a reliable pharmacological tool to serve as an optimizer of a psychedelic experience by inducing positive emotions.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years.
2. Understanding of the German language.
3. Understanding the procedures and the risks that are associated with the study.
4. Participants must be willing to adhere to the protocol and sign the consent form.
5. Participants must be willing to refrain from taking illicit psychoactive substances during the study.
6. Participants must be willing to drink only alcohol-free liquids and no coffee, black or green tea, or energy drink after midnight of the evening before the study session, as well as during the study day.
7. Participants must be willing not to drive a traffic vehicle or to operate machines within 48 h after substance administration.
8. Willing to use effective birth control throughout study participation.
9. Body mass index between 18-29 kg/m2.

Exclusion Criteria:

1. Chronic or acute medical condition
2. Current or previous major psychiatric disorder
3. Psychotic disorder in first-degree relatives, not including psychotic disorders secondary to an apparent medical reason, e.g. brain injury, dementia, or lesions of the brain.
4. Hypertension (SBP>140/90 mmHg) or hypotension (SBP<85 mmHg)
5. Illicit substance use (not including cannabis) more than 20 times or any time within the previous month
6. Pregnant or nursing women.
7. Participation in another clinical trial (currently or within the last 30 days).
8. Use of medications that may interfere with the effects of the study medications.
9. Tobacco smoking (>10 cigarettes/day).
10. Consumption of alcoholic drinks (>15 drinks/week).

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Acute Subjective effects I | through study completion, an average of 18 months
  The Visual Analog Scales (VAS) assesses the intensity and duration of the subjective effect on a scale from 0 - 100 percent with higher scores representing more intense effects. Assessed 12 times on each study day
Acute Subjective effects II | through study completion, an average of 18 months
  The Adjective Mood Rating Scale (AMRS) assesses the occurrence and intensity of 60 moods on a 4-point Likert scale ranging from "not at all" to "extremely".
Acute Subjective effects III | through study completion, an average of 18 months
  5 Dimensions of Altered States of Consciousness (5D-ASC) consisting of 94 items to be rated on a visual analog scale (0-100 mm), with higher values indicating stronger effects.
Acute autonomic effects I (blood pressure) | through study completion, an average of 18 months
  Blood pressure (systolic and diastolic) will be measured with an automatic oscillometric device.
Acute autonomic effects I (heart rate) | through study completion, an average of 18 months
  Heart rate will be measured with an automatic oscillometric device.
Acute autonomic effects III (body temperature) | through study completion, an average of 18 months
  Body temperature will be measured with an ear thermometer.
Acute autonomic effects IV (ECG QT-time) | through study completion, an average of 18 months
  An ECG will be performed twice: once before and once after substance administration.

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of MDMA and metabolites | through study completion, an average of 18 months
  Assessed via blood samples. Findings will be described descriptively.
Time to peak plasma concentration (Tmax) of MDMA and metabolites | through study completion, an average of 18 months
  Assessed via blood samples. Findings will be described descriptively.
Area under the plasma concentration vs. time curve (AUC) of MDMA and metabolites | through study completion, an average of 18 months
  Assessed via blood samples. Findings will be described descriptively.
Elimination half-life values of MDMA and metabolites | through study completion, an average of 18 months
  Assessed via blood samples. Findings will be described descriptively.
Peak plasma concentration (Cmax) of Psilocybin and metabolites | through study completion, an average of 18 months
  Assessed via blood samples. Findings will be described descriptively.
Time to peak plasma concentration (Tmax) of Psilocybin and metabolites | through study completion, an average of 18 months
  Assessed via blood samples. Findings will be described descriptively.
Area under the concentration vs. time curve (AUC) of Psilocybin and metabolites | through study completion, an average of 18 months
  Assessed via blood samples. Findings will be described descriptively.
Elimination half-life values of Psilocybin and metabolites | through study completion, an average of 18 months
  Assessed via blood samples. Findings will be described descriptively.
Plasma concentration of Oxytocin | through study completion, an average of 18 months
  Assessed via blood samples.
States of Consciousness Questionnaire | through study completion, an average of 18 months
  Assesses the emergence and intensity of phenomenons occurring in altered states of consciousness on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely")
Spiritual Realms Questionnaire | through study completion, an average of 18 months
  Assesses the spiritual phenomenons elicited by psychedelic substances through 11 main questions to be answered on a total of 65 sub-ordered 100mm visual analog scales once on each study day
Subacute effects on general and mental well-being I (WEMWBS) | through study completion, an average of 18 months
  The Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) is a 14-item questionnaire, that covers different concepts associated with positive mental health, including both hedonic and eudaimonic aspects, positive affect, satisfying interpersonal relationships and positive functioning. For each item an ordinal five point frequency answer format, ranging from 1 = none of the time" to 5 = "all of the time" is applied.
Subacute effects on general and mental well-being II (GHQ-12) | through study completion, an average of 18 months
  The General Health Questionnaire (GHQ-12) consists of a 12-item questionnaire with a four-point response scale assessing general psychological discomfort.
Subacute effects on general and mental well-being III (SPANE) | through study completion, an average of 18 months
  The Scale of Positive and Negative Experience (SPANE) is a 12-item questionnaire to capture the affective component of subjective well-being. The SPANE includes six items to assess positive feelings and six items to assess negative feelings. The feelings are reported on a 5-point scale ranging from "very rarely" to "very often or always".
Subacute effects on general and mental well-being IV (BFW/E) | through study completion, an average of 18 months
  The "Positive Attitude towards Life" is an 8-item subscale of the 39-item Bern Subjective Well-Being Questionnaire for adults. A six-point rating scale ranging from 1 ('strongly disagree') to 6 ('strongly agree') is used to rate the attitude towards life.
Subacute effects on general and mental well-being V (GLS) | through study completion, an average of 18 months
  Global life satisfaction is assessed based on a single item life satisfaction measure which is a simple, yet widespread approach. The question is answered on a 11-point scale: "In general, how satisfied are you with your life if 0 means 'not at all satisfied' and 10 means 'completely satisfied'?".
Adverse effects (acute and subacute) | through study completion, an average of 18 months
  The 2011 revised Beschwerden-Liste (B-LR) consists of a 40-item list covering a wide variety of symptoms and complaints that are answered with a four-point intensity-scoring ranging from "not at all" to "strong".
Effects on Appreciation | through study completion, an average of 18 months
  The Appreciation Scale (AS) comprises 57 items used to measure aspects of appreciation. Subjects are asked to rate themselves on a scale from 1 to 7 in terms of either attitude intensity ('strongly disagree' to 'strongly agree') or frequency ('never' to 'more than once a day'). Scores on the subscales are summed up to yield a score representing the overall degree of appreciation (or level of appreciativeness), with higher scores indicating more of the positive construct.
Effect moderation by personality traits I (NEO-FFI) | Baseline
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The NEO Five Factor Inventory (NEO-FFI) is a self-description questionnaire with 60 items for the measurement of the "big five": neuroticism, extraversion, openness, agreeableness, and consciousness. It uses a 5-point Likert scale ranging from "completely disagree" to "fully agree".
Effect moderation by personality traits II (FPI-R) | Baseline
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The Freiburger Personality Inventory (FPI-R) version comprises 138 items and covers 12 dimensions of personality: life satisfaction, social orientation, performance orientation, inhibition, excitability, aggressiveness, stress, physical complaints, health concerns, openness, as well as the secondary factors according to Eysenck's Extraversion and Emotionality (Neuroticism). It uses a 2-point scale ("true" and "not true").
Effect moderation by personality traits III (SPF) | Baseline
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The Saarbrücker Persönlichkeitsfragebogen (SPF) defines empathy as the "reactions of one individual to the observed experiences of another." It assesses 28-items on a 5-point Likert scale ranging from "Does not describe me well" to "Describes me very well". The measure has 4 subscales (Perspective Taking, Fantasy, Empathic Concern, Personal Distress) each made up of 7 different items.
Effect moderation by personality traits IV (HEXACO) | Baseline
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The HEXACO personality inventory is a six-dimensional model of human personality with 100 items.The six factors are: Honesty-Humility, Emotionality, Extraversion, Agreeableness, Conscientiousness and Openness to Experience.
Effect moderation by personality traits V (DSQ-40) | Baseline
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The Defense Style Questionnaire (DSQ-40) can provide scores for 20 individual defenses, and scores for the three factors "mature", "neurotic", and "immature". Each item is evaluated on a scale from 1 to 9, where "1" indicates "completely disagree" and "9" indicates "fully agree".

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, Prof. Dr. MD, Principal Investigator — University Hospital Basel, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided